CLINICAL TRIAL: NCT01950910
Title: Establishment of a Tissue Bank (Blood, CSF) for the Understanding of the Disease Progression and Early Diagnosis of Motor Neuron Disease (MND).
Brief Title: Establishment of a Tissue Bank (Blood, CSF) for the Understanding of Motor Neuron Disease (MND)
Acronym: WBC
Status: Terminated | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: CHS-Neurology-WBC Tissue Bank
Record Dates: First submitted 2013-03-30; First posted 2013-09-26 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; motor neuron disease; biological markers; biomarkers
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples (serum and protein/RNA/DNA from blood cells) and CSF
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- subjects w/ non-motor neurodegenerative disease: subjects with ALS or with non-motor neurodegenerative disease
- subjects w/out motorneuron degenerative dis: subjects without motorneuron degenerative disease

SUMMARY:
Biomarkers are essential for the identification of disease states. There are no early diagnostic or prognostic markers for ALS. The purpose of this study is to identify a panel of biomarkers from blood or spinal fluid of ALS patients and to collect data to better understand disease progression.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a motor neuron disease characterized by progressive degeneration of motor neurons, muscle atrophy and paralysis. There is no reliable early diagnostic test for ALS making identification of the disease difficult at its earliest stages. Early detection is critical to the initiation of early neuroprotective therapy. By the time a reliable diagnosis can be made, substantial damage to motor neurons and muscle has already occurred. The purpose of the current project is to establish a bank of blood samples (serum and protein/RNA/DNA from blood cells) and CSF for use in the development of an early diagnostic test for ALS and to better understand the progression of this disease.

Samples from patients that have a confirmed or unknown diagnosis of motor neuron disease will be examined. ALS and suspected neuromuscular disease (control) samples will be collected for comparison. Investigators will examine various biochemical, metabolic and genetic markers from these samples in hopes of finding differences in the expression between control subjects and ALS patients and how these biomarkers vary during disease progression. Participants will be asked to complete an optional questionnaire to collect data including medication and vitamin use and medical and disease history. This data will be linked to the patient's samples; however, all samples will be deidentified and coded to avoid the possibility of linking results to the patient. Results will not be stored in the patient's medical record.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older

Exclusion Criteria:

* less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALS patients in the Charlotte, NC, area.
Sampling Method: Non-Probability Sample
Enrollment: 766 (Actual)
Dates: Start 2004-03-29 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Levels of ALS biomarkers in blood | After blood is collected from study subjects. Data will be analyzed at one year.
  Blood samples will be processed to obtain serum samples and to isolate peripheral blood mononuclear cells (PBMC's). Serum samples will be analyzed for biochemical and metabolic markers of interest and future cell culture as needed. PBMCs will be processed for RNA, DNA or protein isolation. Aliquots of all samples will be stored for future study.
Levels of ALS biomarkers in CSF | After CSF is collected from study subject. Data will be analyzed at one year.
  CSF samples will be processed and assayed for biomarkers of interest. An aliquot of CSF sample will be stored for future study.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin R Brooks, MD, Principal Investigator — Neurosciences Institute, Neurology - Charlotte
Locations (1):
- Neurosciences Institute, Neurology - Charlotte, Charlotte, North Carolina, United States